CLINICAL TRIAL: NCT02771561
Title: PFO Closure for Obstructive Sleep Apnoea-1 Study
Brief Title: PFO Closure for Obstructive Sleep Apnoea
Acronym: PCOSA-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P01725
Record Dates: First submitted 2016-05-05; First posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Patent Foramen Ovale; Obstructive Sleep Apnea
Keywords: Patent Foramen Ovale; Obstructive Sleep Apnea; Apnea-Hypopnea Index; Oxygen Desaturation Index; Epworth Sleepiness Scale; Quality of life; Continuous Positive Airway Pressure; Obstructive Sleep Apnea-Hypopnea Syndrome; Gore™ septal occluder device
MeSH Terms: conditions — Foramen Ovale, Patent; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patent Foramen Ovale Closure (Other): All eligible participants undergo a patent foramen ovale closure procedure
  Interventions: Procedure: Patent Foramen Ovale Closure

INTERVENTIONS:
Procedure: Patent Foramen Ovale Closure — Transoesophageal guided percutaneous patent foramen ovale closure using Gore™ septal occluder device

SUMMARY:
Obstructive sleep apnoea (OSA) is a condition which involves episodes of interrupted breathing during sleep due to repetitive narrowing or collapse of the throat. These episodes are usually associated with a drop in blood oxygen levels and brief awakenings, which disrupt the sleep of those affected and can lead to daytime sleepiness. OSA is associated with an increased risk of heart disease and stroke.

In some individuals, the low oxygen levels in the blood can be made worse by also having a small hole in the heart, called a patent foramen ovale (PFO). This hole is present at birth in everyone, but in some people (about 30% of the normal population) it fails to close. Usually a PFO does not cause any medical problems. However, it may be recommended to have a PFO closed by key-hole surgery if someone suffers a stroke, severe migraine or if they are professional divers. There is a higher incidence of PFO in patients with OSA (25-50%) compared to the wider population and this may account for some of the observed increased risk of heart disease and stroke in patients with OSA.

This study will assess the number of patients with OSA who also have a PFO, and whether closing the PFO can improve the symptoms of OSA (e.g. sleepiness, exercise capacity and general well-being), thereby enabling the patient to not be reliant on treatment for OSA. If the study shows that closing the PFO is beneficial then the investigators will assess in a larger study if this treatment can also reduce heart disease and strokes.

DETAILED DESCRIPTION:
Under normal conditions an interatrial communication allows blood to shunt from left to right due to a higher pressure in the left atrium than the right atrium and a greater compliance of the right ventricle than the left ventricle. Right-to-left interatrial shunting (RLS) is usually associated with spontaneous or induced pulmonary hypertension. RLS may occur spontaneously during a release phase of a Valsalva manoeuvres that transiently generates a right to left pressure gradient across the interatrial septum or rarely due to a condition termed platypnea-orthodeoxia. The latter is characterized by dyspnoea and deoxygenation accompanying a change to a sitting or standing from a recumbent position. Platypnea-orthodeoxia is thought to be due to a combination of an interatrial communication and an anatomical variant e.g. a persistent Eustachian valve and/or stretching and distortion of atrial septum allowing more streaming of venous blood from inferior vena cava through the defect when in the upright position. The recommended treatment of platypnea-orthodeoxia is percutaneous closure of patent foramen ovale (PFO).

Obstructive Sleep Apnoea - Hypopnoea Syndrome (OSAHS) is characterised by repetitive upper airway obstruction during sleep causing apnoea (cessation of breathing) and oxygen desaturation. It is a significant health burden on the National Health Service (NHS) and society, affecting approximately 4% middle aged men and 2% middle-aged women. The risk of OSAHS rises with increasing body weight, active smoking and age. OSAHS is set to reach epidemic proportions as the Western population ages and the incidence of obesity rises. About 1% of men in the United Kingdom (UK) have severe OSAHS with an apnoea-hypopnoea index (AHI; the average number of episodes of apnoeas and hypopnoeas per hour of sleep) of >20 and oxygen desaturation index (ODI; the number of desaturation episodes defined as ≥4% drop in oxygen saturations per hour during sleep) of >20, measured by nocturnal oximetry and respiratory polygraphy (intermediate sleep study or Embletta™). Patients with untreated severe OSAHS have a higher incidence of fatal (OR 2.87) and non-fatal (OR 3.17) cardiovascular events compared to age and sex matched controls. The degree of oxygen desaturation inversely correlates with survival and the link is thought to be multifactorial; raised blood viscosity due to increased haematocrit, sympathetic activation leading to arrhythmias and systemic hypertension are thought to be important. In a Cox model a 1% decrease in average nocturnal oxygen saturation (SaO2) was associated with a 33% increase in the incident risk of fatal and nonfatal cardiovascular events. Treatment with continuous positive airways pressure (CPAP) ventilation at night reduces symptoms (snoring, mood, day time sleepiness and headache) and cardiovascular event rate, but it is poorly tolerated and refused by up to a fifth of patients. Improvement in ODI and sleepiness in OSAHS treated by CPAP is transient and when CPAP is discontinued, measurements return to baseline within 1 week.

PFO is found with a higher incidence in patients with OSAHS than controls (69% vs. 17%) and may exacerbate the oxygen desaturation in OSAHS during apnoeic/ hypopnoeic episodes observed in some patients. In OSAHS patients with greater ODI to AHI ratio (ODI/AHI>0.67), the prevalence of large PFO was nine out of 15 (60%) versus two out of 15 (13%) in those with ODI/AHI <0.33. OSAHS is believed to raise right heart pressures and increase RLS via the interatrial defect due to repeated nocturnal Valsalva and Muller manoeuvres. Prolonged oxygen desaturation may further exacerbate sleep apnoea by decreasing central respiratory drive. In selected populations of OSAHS patients, PFO closure may be beneficial. This has been reported in a number of case reports but has not been studied in a larger trial population.

Hypothesis:

RLS via a PFO in patients with severe OSAHS: ESS≥11 and ODI≥20 or ODI/AHI >0.67, is deleterious and closing the PFO will improve oxygen saturation, exercise tolerance, symptoms, quality of life and will reduce CPAP requirement and, ultimately, will reduce the incidence of fatal/ non-fatal cardiovascular events.

This study will assess the improvement of symptoms of OSA (e.g. sleepiness, exercise capacity and general well-being) following PFO closure. Improving symptoms will enable patients to not be reliant on treatment for OSA. If PFO closure is beneficial the investigator aims to assess the efficacy of treatment to reduce heart disease and strokes in a larger study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Diagnosis of obstructive sleep apnoea-hypopnoea syndrome (OSAHS)
* Epworth Sleepiness Scale score of 11 or greater
* Oxygen Desaturation Index of 20 or greater (and/or oxygen desaturation index/apnoea-hypopnoea index greater than 0.67)
* Naive to Continuous Positive Airway Pressure (CPAP) treatment, or CPAP intolerant (defined at any review as: CPAP use less than 4 hours per night and unable to tolerate/receive no benefit, or at clinical discretion), or poor CPAP responders (defined at any review as: failure to improve Epworth Sleepiness Scale score by more than 4 points from Epworth Sleepiness Scale score at diagnostic visit plus persistent symptoms suggesting poorly controlled OSAHS and/or a prior failure to tolerate CPAP therapy)
* Moderate to large Patent Foramen Ovale (PFO) as seen on a transthoracic echocardiogram bubble study

CPAP naive patients with moderate-large PFO will start CPAP treatment during the study, but outcomes will be assessed at baseline (before starting CPAP treatment) and at six months post PFO closure (after one week of CPAP abstinence).

Exclusion Criteria:

* Coexistent significant respiratory disease (FEV1 <50% predicted)
* Weight >180kg (maximum weight allowance for echocardiogram table)
* Known or suspected pregnancy
* Other cardiac disease (valve disease, known cardiomyopathy, left ventricular failure, known congenital heart disease)
* Previous atrial septal closure device
* Inability to give informed consent or comply with the protocol
* Anatomically unsuitable for percutaneous PFO closure with Gore™ septal occluder device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in Epworth Sleepiness Scale | Change from baseline Epworth Sleepiness Scale score at six months post Patent Foramen Ovale Closure
Change in Apnoea-Hypopnoea Index | Change from baseline Apnoea-Hypopnoea Index at six months post Patent Foramen Ovale Closure
Change in Oxygen Desaturation Index | Change from baseline Oxygen Desaturation Index at six months post Patent Foramen Ovale Closure
Change in Six Minute Walk Test | Change from baseline six minute walk test at six months post Patent Foramen Ovale Closure
Change in Sleep Apnea Quality of Life Index (SAQLI) | Change from baseline SAQLI at six months post Patent Foramen Ovale Closure
Change in Functional Outcomes of Sleep Questionnaire (FOSQ) | Change from baseline FOSQ at six months post Patent Foramen Ovale Closure
Change in Short Form (36) Health Survey (SF36) | Change from baseline SF36 at six months post Patent Foramen Ovale Closure

SECONDARY OUTCOMES:
Change in Continuous Positive Airway Pressure (CPAP) | Change from baseline CPAP use at six months post Patent Foramen Ovale Closure
  CPAP use = the hours of use per 24 hour period. This is recorded by the CPAP device.
Cardiovascular events (CV) | Six months post Patent Foramen Ovale Closure
  Incidence of fatal and non-fatal CV events

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Hoole, BM BCh, Principal Investigator — Papworth Hospital NHS Foundation Trust; Michael Davies, MB BS, Principal Investigator — Papworth Hospital NHS Foundation Trust
Locations (1):
- Papworth Hospital NHS Foundation Trust, Papworth Everard, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We do not plan to make individual participant data available.

REFERENCES:
- [Background] Agnoletti G, Iserin L, Lafont A, Sidi D, Desnos M. Obstructive sleep apnoea and patent foramen ovale: successful treatment of symptoms by percutaneous foramen ovale closure. J Interv Cardiol. 2005 Oct;18(5):393-5. doi: 10.1111/j.1540-8183.2005.00072.x. PMID 16202118
- [Background] Beelke M, Angeli S, Del Sette M, De Carli F, Canovaro P, Nobili L, Ferrillo F. Obstructive sleep apnea can be provocative for right-to-left shunting through a patent foramen ovale. Sleep. 2002 Dec;25(8):856-62. PMID 12489891
- [Background] Bradley TD, Martinez D, Rutherford R, Lue F, Grossman RF, Moldofsky H, Zamel N, Phillipson EA. Physiological determinants of nocturnal arterial oxygenation in patients with obstructive sleep apnea. J Appl Physiol (1985). 1985 Nov;59(5):1364-8. doi: 10.1152/jappl.1985.59.5.1364. PMID 4066566
- [Background] Engleman HM, Martin SE, Kingshott RN, Mackay TW, Deary IJ, Douglas NJ. Randomised placebo controlled trial of daytime function after continuous positive airway pressure (CPAP) therapy for the sleep apnoea/hypopnoea syndrome. Thorax. 1998 May;53(5):341-5. doi: 10.1136/thx.53.5.341. PMID 9708223
- [Background] Johansson MC, Eriksson P, Peker Y, Hedner J, Rastam L, Lindblad U. The influence of patent foramen ovale on oxygen desaturation in obstructive sleep apnoea. Eur Respir J. 2007 Jan;29(1):149-55. doi: 10.1183/09031936.00035906. Epub 2006 Sep 27. PMID 17005584
- [Background] La Rovere MT, Pinna GD, Hohnloser SH, Marcus FI, Mortara A, Nohara R, Bigger JT Jr, Camm AJ, Schwartz PJ; ATRAMI Investigators. Autonomic Tone and Reflexes After Myocardial Infarcton. Baroreflex sensitivity and heart rate variability in the identification of patients at risk for life-threatening arrhythmias: implications for clinical trials. Circulation. 2001 Apr 24;103(16):2072-7. doi: 10.1161/01.cir.103.16.2072. PMID 11319197
- [Background] Marin JM, Carrizo SJ, Vicente E, Agusti AG. Long-term cardiovascular outcomes in men with obstructive sleep apnoea-hypopnoea with or without treatment with continuous positive airway pressure: an observational study. Lancet. 2005 Mar 19-25;365(9464):1046-53. doi: 10.1016/S0140-6736(05)71141-7. PMID 15781100
- [Background] Shanoudy H, Soliman A, Raggi P, Liu JW, Russell DC, Jarmukli NF. Prevalence of patent foramen ovale and its contribution to hypoxemia in patients with obstructive sleep apnea. Chest. 1998 Jan;113(1):91-6. doi: 10.1378/chest.113.1.91. PMID 9440574
- [Background] Silver B, Greenbaum A, McCarthy S. Improvement in sleep apnea associated with closure of a patent foramen ovale. J Clin Sleep Med. 2007 Apr 15;3(3):295-6. PMID 17561600
- [Background] Smith ML, Niedermaier ON, Hardy SM, Decker MJ, Strohl KP. Role of hypoxemia in sleep apnea-induced sympathoexcitation. J Auton Nerv Syst. 1996 Jan 5;56(3):184-90. doi: 10.1016/0165-1838(95)00062-3. PMID 8847442
- [Background] van den Aardweg JG, Karemaker JM. Repetitive apneas induce periodic hypertension in normal subjects through hypoxia. J Appl Physiol (1985). 1992 Mar;72(3):821-7. doi: 10.1152/jappl.1992.72.3.821. PMID 1568978
- [Background] Young T, Palta M, Dempsey J, Peppard PE, Nieto FJ, Hla KM. Burden of sleep apnea: rationale, design, and major findings of the Wisconsin Sleep Cohort study. WMJ. 2009 Aug;108(5):246-9. PMID 19743755
- [Background] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434
- [Background] Zoccali C, Mallamaci F, Tripepi G. Nocturnal hypoxemia predicts incident cardiovascular complications in dialysis patients. J Am Soc Nephrol. 2002 Mar;13(3):729-733. doi: 10.1681/ASN.V133729. PMID 11856778